CLINICAL TRIAL: NCT00976599
Title: An Exploratory Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study To Assess The Pharmacodynamics Of CP-690,550, Administered Orally Twice Daily (BID) For 4 Weeks, In Subjects With Active Rheumatoid Arthritis
Brief Title: A Study To Evaluate The Mechanism Of Action Of CP-690,550 In Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: A3921073
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2012-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CP-690,550 + methotrexate (Experimental)
  Interventions: Drug: CP-690,550 + methotrexate
- Placebo + methotrexate (Placebo Comparator)
  Interventions: Drug: Placebo + Methotrexate

INTERVENTIONS:
Drug: CP-690,550 + methotrexate — CP-690,550 dose is 10 mg twice daily, oral tablets, for 4 weeks Methotrexate dose is ≥ 7.5 mg / week and ≤ 25 mg / week
  Arms: CP-690,550 + methotrexate
Drug: Placebo + Methotrexate — Methotrexate dose is ≥ 7.5 mg / week and ≤ 25 mg / week
  Arms: Placebo + methotrexate

SUMMARY:
To explore the effect of CP-690,550 on blood and synovial markers in subjects with rheumatoid arthritis. To evaluate the safety, tolerability and efficacy of CP-690,550.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a diagnosis of rheumatoid arthritis based on the American College of Rheumatology Association
* The subject has active disease at both Screening and Baseline, as defined:

  * ≥4 joints tender or painful on motion, AND
  * ≥4 joints swollen;
* The subject must have at least one knee, one elbow, one wrist or two metacarpophalangeal joints with active synovitis suitable for biopsy by the shaver technique

Exclusion Criteria:

* No arthroscopy should have been performed in the past 3 months in the same joint that is to be biopsied in this study.
* No intra-articular steroids should have been injected in the joint to be biopsied in this study in the previous 3 months.
* Subjects with evidence of hematopoietic disorders or evidence of hemoglobin levels < 9.0 gm/dL or hematocrit < 30 % at screening visit or within the 3 months prior to baseline synovial biopsy.
* An absolute white blood cell (WBC) count of < 3.0 x 109/L (<3000/mm3) or absolute neutrophil count of <1.2 X 109/L (<1200/mm3) at screening visit or within the 3 months prior to baseline synovial biopsy.
* Thrombocytopenia, as defined by a platelet count <100 x 109/L (< 100,000/mm3) at screening visit or within the 3 months prior to baseline synovial biopsy.
* Estimated GFR less than 40 ml/min based on Cockcroft Gault calculation .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (11):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Battle Creek, Michigan
  - Pfizer Investigational Site, Mayfield Village, Ohio
  - Pfizer Investigational Site, Mentor, Ohio
  - Pfizer Investigational Site, Willoughby, Ohio
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Mesquite, Texas
  - Pfizer Investigational Site, Sunnyvale, Texas
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Hetland ML, Strangfeld A, Bonfanti G, Soudis D, Deuring JJ, Edwards RA. Machine learning prediction and explanatory models of serious infections in patients with rheumatoid arthritis treated with tofacitinib. Arthritis Res Ther. 2024 Aug 27;26(1):153. doi: 10.1186/s13075-024-03376-9. PMID 39192350
- [Derived] Wright GC, Mysler E, Kwok K, Cadatal MJ, Germino R, Yndestad A, Kinch CD, Ogdie A. Impact of Race on the Efficacy and Safety of Tofacitinib in Rheumatoid Arthritis: Post Hoc Analysis of Pooled Clinical Trials. Rheumatol Ther. 2024 Oct;11(5):1135-1164. doi: 10.1007/s40744-024-00677-y. Epub 2024 Jul 3. PMID 38958913
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Hansen KE, Mortezavi M, Nagy E, Wang C, Connell CA, Radi Z, Litman HJ, Adami G, Rossini M. Fracture in clinical studies of tofacitinib in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2022 Dec 27;14:1759720X221142346. doi: 10.1177/1759720X221142346. eCollection 2022. PMID 36601090
- [Derived] Curtis JR, Yamaoka K, Chen YH, Bhatt DL, Gunay LM, Sugiyama N, Connell CA, Wang C, Wu J, Menon S, Vranic I, Gomez-Reino JJ. Malignancy risk with tofacitinib versus TNF inhibitors in rheumatoid arthritis: results from the open-label, randomised controlled ORAL Surveillance trial. Ann Rheum Dis. 2023 Mar;82(3):331-343. doi: 10.1136/ard-2022-222543. Epub 2022 Dec 5. PMID 36600185
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Wang L, Chen C, Kwok K, Biswas P, Shapiro A, Madsen A, Wollenhaupt J. Long-term safety of tofacitinib up to 9.5 years: a comprehensive integrated analysis of the rheumatoid arthritis clinical development programme. RMD Open. 2020 Oct;6(3):e001395. doi: 10.1136/rmdopen-2020-001395. PMID 33127856
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Cohen SB, Tanaka Y, Mariette X, Curtis JR, Lee EB, Nash P, Winthrop KL, Charles-Schoeman C, Thirunavukkarasu K, DeMasi R, Geier J, Kwok K, Wang L, Riese R, Wollenhaupt J. Long-term safety of tofacitinib for the treatment of rheumatoid arthritis up to 8.5 years: integrated analysis of data from the global clinical trials. Ann Rheum Dis. 2017 Jul;76(7):1253-1262. doi: 10.1136/annrheumdis-2016-210457. Epub 2017 Jan 31. PMID 28143815
- [Derived] Boyle DL, Soma K, Hodge J, Kavanaugh A, Mandel D, Mease P, Shurmur R, Singhal AK, Wei N, Rosengren S, Kaplan I, Krishnaswami S, Luo Z, Bradley J, Firestein GS. The JAK inhibitor tofacitinib suppresses synovial JAK1-STAT signalling in rheumatoid arthritis. Ann Rheum Dis. 2015 Jun;74(6):1311-6. doi: 10.1136/annrheumdis-2014-206028. Epub 2014 Nov 14. PMID 25398374
- [Derived] Cohen S, Radominski SC, Gomez-Reino JJ, Wang L, Krishnaswami S, Wood SP, Soma K, Nduaka CI, Kwok K, Valdez H, Benda B, Riese R. Analysis of infections and all-cause mortality in phase II, phase III, and long-term extension studies of tofacitinib in patients with rheumatoid arthritis. Arthritis Rheumatol. 2014 Nov;66(11):2924-37. doi: 10.1002/art.38779. PMID 25047021
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921073&StudyName=A%20Study%20To%20Evaluate%20The%20Mechanism%20Of%20Action%20Of%20CP-690%2C550%20In%20Patients%20With%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550: CP-690,550 10 milligram (mg) tablet orally twice daily up to Day 27 followed by single oral dose on Day 28.
- Placebo: Placebo matched to CP-690,550 10 mg tablet orally twice daily up to Day 27 followed by single oral dose on Day 28.
Period: Overall Study
Arm/Group | CP-690,550 | Placebo
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CP-690,550: CP-690,550 10 mg tablet orally twice daily up to Day 27 followed by single oral dose on Day 28.
- Total: Total of all reporting groups
Arm/Group | CP-690,550 | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.2) | 53.1 (14.3) | 53.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Synovial Tissue Messenger Ribonucleic Acid (mRNA) Expression at Day 28
Description: Synovial tissue biopsy were performed and assayed for mRNA gene expression by quantitative polymerized chain reaction (PCR) using standard curve method. Standard curve generated by linear regression using log threshold cycle versus log (cell number). Interleukin-1beta (IL-1beta), IL-6, matrix metalloproteinase-3 (MMP3), cluster of differentiation 19 (CD19), cluster of differentiation 3 epsilon (CD3E), Janus kinase 1 (JAK1), JAK2, JAK3, signal transducers, activators of transcription (STAT1), interferon stimulated gene 15 (ISG15), C-X-C motif chemokine 10 (CXCL10), chemokine (C-C motif) ligand2 (CCL2), phospho-STAT1 (pSTAT1), pSTAT3, tumor necrosis factor alpha (TNFalpha), receptor activator of nuclear factor kappa-B ligand (RANKL) and osteoprotegerin (OPG) presented as control gene normalized expression (relative expression) within synovial tissue.
Time Frame: Day -7 (Baseline), Day 28
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of the study medication. Analyses of tumor necrosis factor alpha(TNFα), receptor activator of nuclear factor kappa-B ligand(RANKL), osteoprotegerin(OPG) were not performed due to insufficient samples and lack of appropriate method to process/analyze samples.
Measure: Mean (Standard Deviation); unit: relative expression unit (REU)
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
relative expression unit (REU)
  Baseline: IL-1beta mRNA | -2.73 (0.77) | -2.83 (0.80)
  Baseline: IL-6 mRNA | -3.72 (0.67) | -3.96 (0.55)
  Baseline: MMP3 mRNA | -2.01 (1.39) | -2.52 (1.64)
  Baseline: CD19 mRNA | -2.98 (1.25) | -3.46 (1.34)
  Baseline: CD3E mRNA | -1.58 (0.71) | -1.75 (0.58)
  Baseline: JAK1 mRNA | 0.30 (0.24) | 0.31 (0.29)
  Baseline: JAK2 mRNA | 0.17 (0.26) | 0.15 (0.25)
  Baseline: JAK3 mRNA | -0.77 (0.40) | -0.88 (0.52)
  Baseline: STAT1 mRNA | -0.43 (0.29) | -0.46 (0.33)
  Baseline: ISG15 mRNA | -1.26 (0.23) | -1.33 (0.27)
  Baseline: CXCL10 mRNA | -1.21 (0.85) | -1.24 (0.81)
  Baseline: CCL2 mRNA | -1.70 (0.29) | -1.73 (0.39)
  Baseline: pSTAT1 protein | 0.18 (0.33) | 0.27 (0.39)
  Baseline: pSTAT3 protein | 0.77 (0.29) | 0.79 (0.30)
  Change at Day 28: IL-1beta mRNA | -0.01 (0.88) | 0.09 (0.43)
  Change at Day 28: IL-6 mRNA | -0.25 (0.86) | -0.08 (0.45)
  Change at Day 28: MMP3 mRNA | -0.80 (0.92) | -0.03 (1.23)
  Change at Day 28: CD19 mRNA | 0.06 (0.85) | -0.31 (0.72)
  Change at Day 28: CD3E mRNA | -0.07 (0.53) | -0.12 (0.44)
  Change at Day 28: JAK1 mRNA | 0.04 (0.36) | -0.10 (0.36)
  Change at Day 28: JAK2 mRNA | -0.07 (0.40) | -0.10 (0.29)
  Change at Day 28: JAK3 mRNA | -0.05 (0.35) | -0.13 (0.52)
  Change at Day 28: STAT1 mRNA | -0.15 (0.46) | 0.01 (0.35)
  Change at Day 28: ISG15 mRNA | -0.16 (0.40) | 0.11 (0.34)
  Change at Day 28: CXCL10 mRNA | -0.49 (0.75) | 0.15 (0.61)
  Change at Day 28: CCL2 mRNA | -0.20 (0.30) | -0.02 (0.28)
  Change at Day 28: pSTAT1 protein | -0.20 (0.44) | -0.10 (0.36)
  Change at Day 28: pSTAT3 protein | -0.10 (0.42) | -0.10 (0.18)

2. Primary Outcome: Change From Baseline in Protein Expression of Tumor Necrosis Factor Alpha (TNFalpha), Interleukin-6 (IL-6), Interleukin-17a (IL-17a) and Interleukin-10 (IL-10) at Day 28
Description: Synovial tissue biopsy was to be performed and assayed for protein expression by quantitative PCR using standard curve method. Standard curve was to be generated by linear regression using log threshold cycle versus log (cell number). TNFalpha, IL-6, IL-17 and IL-10 data were to be presented as control normalized expression (relative expression) within synovial tissue.
Time Frame: Baseline (Day -7), Day 28
Population: Analyses of TNFalpha, IL-6, IL-17 and IL-10 were not performed due to insufficient samples and lack of appropriate method to process/analyze the samples.
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change From Baseline in Percentage of Area Stained For CD3+ and CD68+ Surface Markers of Inflammatory Cells of the Synovial Tissue at Day 28
Description: The intensity of CD3 and CD68 cell infiltration was expressed as the percentage area of the tissue section occupied by positively stained cells. Surface marker CD68 macrophages and CD3 thymus cells (T cells) in the inflammatory cells of synovial tissue were detected by immunohistochemical staining.
Time Frame: Baseline (Day -7), Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure. n=number of participants evaluable at specific time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: percentage area stained
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 12 | 12
percentage area stained
  Baseline: CD3+ Cells (n=12, 12) | 7.33 (6.12) | 7.92 (7.49)
  Baseline: CD68+ Cells (n=12, 13) | 31.83 (20.59) | 32.85 (26.05)
  Change at Day 28: CD3+ Cells (n=10, 8) | 1.50 (3.95) | 0.13 (7.38)
  Change at Day 28: CD68+ Cells (n=12, 11) | 1.67 (19.86) | 0.82 (18.37)

4. Primary Outcome: Blood Levels for Gene Expression (Messenger Ribonucleic Acid [mRNA]) at Baseline (Day-7)
Description: Blood levels were utilized for expression analysis (mRNA) of following genes that reflect immune function: CD19, CD3 epsilon (CD3E), STAT1, STAT3, ISG15, CXCL10. mRNA gene expression in blood were assayed by quantitative PCR using standard curve method. Standard curve generated by linear regression using log threshold cycle versus log (cell number). Data were presented as control gene normalized expression (relative expression) within blood.
Time Frame: Baseline (Day -7)
Population: FAS included all randomized participants who received at least 1 dose of the study medication. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: REU
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
REU
  CD19 mRNA | 0.11 (0.28) | 0.29 (0.25)
  CD3E mRNA | 0.41 (0.44) | 0.40 (0.38)
  STAT1 mRNA | 0.06 (0.25) | 0.02 (0.13)
  STAT3 mRNA | 0.61 (0.13) | 0.64 (0.08)
  ISG15 mRNA | -0.65 (0.45) | -0.56 (0.47)
  CXCL10 mRNA | -1.58 (0.33) | -1.65 (0.19)

5. Primary Outcome: Blood Levels for Gene Expression (Messenger Ribonucleic Acid [mRNA]) at Day 28
Description: Blood levels were utilized for expression analysis (mRNA) of following genes that reflect immune function: CD19, CD3E, STAT1, STAT3, ISG15, CXCL10. mRNA gene expression in blood were assayed by quantitative PCR using standard curve method. Standard curve generated by linear regression using log threshold cycle versus log (cell number). Data were presented as control gene normalized expression (relative expression) within blood.
Time Frame: Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: REU
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
REU
  CD19 mRNA | 0.35 (0.24) | 0.30 (0.25)
  CD3E mRNA | 0.49 (0.34) | 0.40 (0.32)
  STAT1 mRNA | -0.01 (0.28) | 0.04 (0.21)
  STAT3 mRNA | 0.60 (0.13) | 0.59 (0.13)
  ISG15 mRNA | -0.93 (0.20) | -0.48 (0.51)
  CXCL10 mRNA | -1.64 (0.22) | -1.59 (0.28)

6. Primary Outcome: Blood Cytokine Level at Pre-dose on Day 1
Description: Blood samples were collected from all the participants and pro-inflammatory cytokine levels were measured. The levels of pro-inflammatory cytokine IL-1beta, IL-1alpha, IL-4, IL-6, IL-8, IL-10, IL-17A, IL-7, IL-21, active 70 kDa (p70) form of IL-12(IL-12p70), interferon gamma (IFNgamma) - induced protein 10 (IP-10), TNFalpha, granulocyte macrophage colony-stimulating factor (GM-CSF), macrophage inflammatory protein 1 alpha (MIP1a), monocyte chemotactic protein 1 (MCP1), soluble vascular endothelial growth factor (sVEGF), soluble vascular cell adhesion molecule 1 (sVCAM-1), soluble intercellular adhesion molecule 1 (sICAM-1), granulocyte colony-stimulating factor (G-CSF) was measured by immunoassay and the levels were expresses as picogram per milliliter (pg/mL).
Time Frame: Pre-dose on Day 1
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL
  IL-1alpha | 0.75 (0.68) | 0.67 (0.68)
  IL-1beta | 0.42 (0.39) | 0.41 (0.41)
  IL-4 | 0.29 (0.29) | 0.17 (0.16)
  IL-6 | 0.97 (0.67) | 0.77 (0.45)
  IL-7 | 0.89 (0.32) | 0.74 (0.23)
  IL-8 | 1.17 (0.24) | 1.19 (0.27)
  IL-10 | 0.25 (0.24) | 0.33 (0.37)
  IL-12p70 | 0.31 (0.29) | 0.35 (0.44)
  IL-17A | 0.49 (0.48) | 0.44 (0.37)
  IL-21 | 1.56 (1.10) | 1.47 (1.04)
  IP-10 | 2.22 (0.23) | 2.23 (0.30)
  TNFalpha | 0.45 (0.43) | 0.44 (0.51)
  IFNgamma | 0.15 (0.16) | 0.11 (0.07)
  G-CSF | 0.57 (0.47) | 0.60 (0.34)
  GM-CSF | 0.48 (0.48) | 0.36 (0.46)
  MCP1 | 2.14 (0.26) | 2.09 (0.32)
  MIP1a | 0.85 (0.45) | 0.90 (0.32)
  sVEGF | 1.96 (0.44) | 1.87 (0.28)
  sVCAM-1 | 4.95 (0.17) | 5.07 (0.17)
  sICAM-1 | 4.65 (0.12) | 4.76 (0.17)

7. Primary Outcome: Blood Cytokine Level at 1 Hour Post-dose on Day 1
Description: Blood samples were collected from all the participants and pro-inflammatory cytokine levels were measured. The levels of pro-inflammatory cytokine IL-1beta, IL-1alpha, IL-4, IL-6, IL-8, IL-10, IL-17A, IL-7, IL-21, IL-12p70, IP-10, TNFalpha, IFNgamma, GM-CSF, MIP1a, MCP1, sVEGF, sVCAM-1, sICAM-1, G-CSF was measured by immunoassay and the levels were expresses as pg/mL.
Time Frame: 1 hour post-dose on Day 1
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL
  IL-1alpha | 0.76 (0.68) | 0.73 (0.68)
  IL-1beta | 0.43 (0.42) | 0.40 (0.43)
  IL-4 | 0.29 (0.28) | 0.15 (0.13)
  IL-6 | 0.90 (0.52) | 0.78 (0.43)
  IL-7 | 0.86 (0.36) | 0.72 (0.26)
  IL-8 | 1.12 (0.31) | 1.15 (0.23)
  IL-10 | 0.23 (0.22) | 0.31 (0.35)
  IL-12p70 | 0.36 (0.31) | 0.34 (0.43)
  IL-17A | 0.58 (0.46) | 0.42 (0.36)
  IL-21 | 1.45 (1.16) | 1.45 (1.07)
  IP-10 | 2.17 (0.25) | 2.22 (0.31)
  TNFalpha | 0.41 (0.46) | 0.44 (0.52)
  IFNgamma | 0.12 (0.07) | 0.10 (0.00)
  G-CSF | 0.56 (0.47) | 0.62 (0.36)
  GM-CSF | 0.49 (0.49) | 0.39 (0.49)
  MCP1 | 2.09 (0.26) | 2.03 (0.33)
  MIP1a | 0.83 (0.47) | 0.89 (0.33)
  sVEGF | 1.98 (0.42) | 1.87 (0.27)
  sVCAM-1 | 4.94 (0.15) | 5.06 (0.17)
  sICAM-1 | 4.64 (0.13) | 4.76 (0.18)

8. Primary Outcome: Blood Cytokine Level at 4 Hours Post-dose on Day 1
Description: as for outcome 7
Time Frame: 4 hours post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
pg/mL
  IL-1alpha | 0.77 (0.69) | 0.65 (0.70)
  IL-1beta | 0.43 (0.46) | 0.41 (0.42)
  IL-4 | 0.28 (0.28) | 0.18 (0.17)
  IL-6 | 0.74 (0.41) | 0.72 (0.39)
  IL-7 | 0.82 (0.39) | 0.73 (0.28)
  IL-8 | 1.18 (0.22) | 1.15 (0.25)
  IL-10 | 0.19 (0.20) | 0.30 (0.35)
  IL-12p70 | 0.35 (0.29) | 0.38 (0.43)
  IL-17A | 0.53 (0.47) | 0.39 (0.40)
  IL-21 | 1.60 (1.09) | 1.36 (1.07)
  IP-10 | 2.10 (0.22) | 2.20 (0.33)
  TNFalpha | 0.41 (0.47) | 0.45 (0.51)
  IFNgamma | 0.17 (0.13) | 0.12 (0.07)
  G-CSF | 0.55 (0.47) | 0.62 (0.41)
  GM-CSF | 0.50 (0.48) | 0.38 (0.48)
  MCP1 | 1.98 (0.29) | 2.07 (0.34)
  MIP1a | 0.81 (0.47) | 0.86 (0.33)
  sVEGF | 1.93 (0.42) | 1.85 (0.28)
  sVCAM-1 | 4.96 (0.15) | 5.03 (0.21)
  sICAM-1 | 4.66 (0.12) | 4.74 (0.20)

9. Primary Outcome: Blood Cytokine Level at Pre-dose on Day 10
Description: as for outcome 7
Time Frame: Pre-dose on Day 10
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL
  IL-1alpha | 0.74 (0.66) | 0.69 (0.68)
  IL-1beta | 0.36 (0.46) | 0.42 (0.43)
  IL-4 | 0.28 (0.28) | 0.19 (0.18)
  IL-6 | 0.68 (0.55) | 0.78 (0.45)
  IL-7 | 0.83 (0.31) | 0.61 (0.38)
  IL-8 | 1.15 (0.29) | 1.21 (0.29)
  IL-10 | 0.21 (0.23) | 0.32 (0.35)
  IL-12p70 | 0.34 (0.32) | 0.34 (0.43)
  IL-17A | 0.50 (0.48) | 0.41 (0.36)
  IL-21 | 1.62 (1.02) | 1.63 (0.86)
  IP-10 | 2.01 (0.25) | 2.18 (0.33)
  TNFalpha | 0.48 (0.49) | 0.48 (0.50)
  IFNgamma | 0.11 (0.05) | 0.11 (0.03)
  G-CSF | 0.60 (0.43) | 0.60 (0.31)
  GM-CSF | 0.48 (0.46) | 0.37 (0.48)
  MCP1 | 2.17 (0.34) | 2.09 (0.38)
  MIP1a | 0.83 (0.52) | 0.89 (0.35)
  sVEGF | 1.93 (0.44) | 1.90 (0.28)
  sVCAM-1 | 4.90 (0.16) | 5.03 (0.16)
  sICAM-1 | 4.63 (0.11) | 4.74 (0.20)

10. Primary Outcome: Blood Cytokine Level at Pre-dose on Day 28
Description: as for outcome 7
Time Frame: Pre-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL
  IL-1alpha | 0.69 (0.71) | 0.68 (0.68)
  IL-1beta | 0.41 (0.45) | 0.39 (0.39)
  IL-4 | 0.24 (0.25) | 0.15 (0.15)
  IL-6 | 0.64 (0.42) | 0.78 (0.32)
  IL-7 | 0.75 (0.34) | 0.53 (0.30)
  IL-8 | 1.19 (0.36) | 1.14 (0.32)
  IL-10 | 0.18 (0.17) | 0.32 (0.31)
  IL-12p70 | 0.27 (0.26) | 0.35 (0.43)
  IL-17A | 0.49 (0.47) | 0.37 (0.37)
  IL-21 | 1.47 (1.08) | 1.53 (0.99)
  IP-10 | 2.01 (0.19) | 2.24 (0.40)
  TNFalpha | 0.46 (0.49) | 0.43 (0.48)
  IFNgamma | 0.11 (0.03) | 0.10 (0.00)
  G-CSF | 0.65 (0.39) | 0.66 (0.34)
  GM-CSF | 0.48 (0.48) | 0.35 (0.45)
  MCP1 | 2.21 (0.35) | 2.09 (0.40)
  MIP1a | 0.84 (0.44) | 0.83 (0.34)
  sVEGF | 1.89 (0.41) | 1.83 (0.27)
  sVCAM-1 | 4.89 (0.14) | 5.01 (0.19)
  sICAM-1 | 4.61 (0.09) | 4.70 (0.21)

11. Primary Outcome: Blood Cytokine Level at 1 Hour Post-dose on Day 28
Description: as for outcome 7
Time Frame: 1 Hour Post-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL
  IL-1alpha | 0.69 (0.68) | 0.69 (0.67)
  IL-1beta | 0.40 (0.41) | 0.39 (0.38)
  IL-4 | 0.25 (0.25) | 0.15 (0.14)
  IL-6 | 0.67 (0.52) | 0.77 (0.39)
  IL-7 | 0.69 (0.38) | 0.61 (0.33)
  IL-8 | 1.10 (0.23) | 1.12 (0.33)
  IL-10 | 0.18 (0.16) | 0.33 (0.33)
  IL-12p70 | 0.33 (0.28) | 0.36 (0.44)
  IL-17A | 0.44 (0.45) | 0.36 (0.34)
  IL-21 | 1.46 (1.06) | 1.52 (0.99)
  IP-10 | 2.00 (0.21) | 2.23 (0.39)
  TNFalpha | 0.39 (0.46) | 0.43 (0.48)
  IFNgamma | 0.12 (0.06) | 0.11 (0.04)
  G-CSF | 0.63 (0.39) | 0.66 (0.29)
  GM-CSF | 0.47 (0.47) | 0.36 (0.45)
  MCP1 | 2.23 (0.30) | 2.06 (0.35)
  MIP1a | 0.81 (0.45) | 0.83 (0.33)
  sVEGF | 1.85 (0.38) | 1.81 (0.26)
  sVCAM-1 | 4.85 (0.15) | 5.04 (0.17)
  sICAM-1 | 4.58 (0.10) | 4.73 (0.23)

12. Primary Outcome: Blood Cytokine Level at 4 Hours Post-dose on Day 28
Description: as for outcome 7
Time Frame: 4 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 13
pg/mL
  IL-1alpha | 0.67 (0.69) | 0.75 (0.66)
  IL-1beta | 0.27 (0.32) | 0.33 (0.39)
  IL-4 | 0.22 (0.27) | 0.14 (0.11)
  IL-6 | 0.56 (0.30) | 0.69 (0.29)
  IL-7 | 0.66 (0.45) | 0.56 (0.36)
  IL-8 | 1.07 (0.21) | 1.07 (0.25)
  IL-10 | 0.16 (0.13) | 0.28 (0.32)
  IL-12p70 | 0.26 (0.27) | 0.31 (0.44)
  IL-17A | 0.37 (0.44) | 0.34 (0.37)
  IL-21 | 1.51 (1.05) | 1.68 (0.92)
  IP-10 | 1.89 (0.21) | 2.13 (0.36)
  TNFalpha | 0.38 (0.42) | 0.38 (0.49)
  IFNgamma | 0.12 (0.07) | 0.11 (0.04)
  G-CSF | 0.57 (0.43) | 0.72 (0.26)
  GM-CSF | 0.49 (0.47) | 0.38 (0.46)
  MCP1 | 2.09 (0.23) | 1.99 (0.38)
  MIP1a | 0.71 (0.48) | 0.80 (0.31)
  sVEGF | 1.80 (0.36) | 1.84 (0.28)
  sVCAM-1 | 4.91 (0.15) | 5.00 (0.14)
  sICAM-1 | 4.61 (0.09) | 4.71 (0.22)

13. Primary Outcome: Blood Cytokine Level at 8 Hours Post-dose on Day 28
Description: as for outcome 7
Time Frame: 8 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 12
pg/mL
  IL-1alpha | 0.76 (0.68) | 0.63 (0.69)
  IL-1beta | 0.29 (0.35) | 0.34 (0.39)
  IL-4 | 0.23 (0.27) | 0.14 (0.12)
  IL-6 | 0.71 (0.39) | 0.79 (0.34)
  IL-7 | 0.67 (0.40) | 0.66 (0.31)
  IL-8 | 1.10 (0.21) | 1.17 (0.26)
  IL-10 | 0.15 (0.11) | 0.29 (0.30)
  IL-12p70 | 0.28 (0.28) | 0.33 (0.42)
  IL-17A | 0.44 (0.42) | 0.29 (0.36)
  IL-21 | 1.58 (1.04) | 1.30 (1.13)
  IP-10 | 1.85 (0.22) | 2.14 (0.35)
  TNFalpha | 0.36 (0.43) | 0.35 (0.48)
  IFNgamma | 0.10 (0.00) | 0.12 (0.07)
  G-CSF | 0.65 (0.37) | 0.83 (0.28)
  GM-CSF | 0.48 (0.45) | 0.38 (0.46)
  MCP1 | 2.11 (0.31) | 2.02 (0.40)
  MIP1a | 0.71 (0.45) | 0.71 (0.35)
  sVEGF | 1.71 (0.36) | 1.82 (0.25)
  sVCAM-1 | 4.87 (0.16) | 5.05 (0.15)
  sICAM-1 | 4.59 (0.09) | 4.74 (0.24)

14. Primary Outcome: Blood Cytokine Level at 24 Hours Post-dose on Day 28
Description: as for outcome 7
Time Frame: 24 Hours Post-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL
  IL-1alpha | 0.73 (0.66) | 0.66 (0.64)
  IL-1beta | 0.38 (0.41) | 0.38 (0.41)
  IL-4 | 0.26 (0.27) | 0.15 (0.15)
  IL-6 | 0.93 (0.42) | 0.99 (0.47)
  IL-7 | 0.79 (0.35) | 0.64 (0.31)
  IL-8 | 1.21 (0.32) | 1.18 (0.29)
  IL-10 | 0.22 (0.17) | 0.30 (0.33)
  IL-12p70 | 0.25 (0.25) | 0.37 (0.44)
  IL-17A | 0.44 (0.44) | 0.32 (0.32)
  IL-21 | 1.54 (0.98) | 1.64 (0.87)
  IP-10 | 2.02 (0.31) | 2.27 (0.39)
  TNFalpha | 0.42 (0.47) | 0.42 (0.51)
  IFNgamma | 0.16 (0.19) | 0.10 (0.00)
  G-CSF | 0.67 (0.39) | 0.71 (0.28)
  GM-CSF | 0.46 (0.46) | 0.31 (0.44)
  MCP1 | 2.33 (0.24) | 2.10 (0.35)
  MIP1a | 0.86 (0.49) | 0.88 (0.28)
  sVEGF | 1.89 (0.41) | 1.84 (0.23)
  sVCAM-1 | 4.88 (0.14) | 5.06 (0.17)
  sICAM-1 | 4.58 (0.10) | 4.74 (0.21)

15. Primary Outcome: Blood Cytokine Level at Pre-dose on Day 35 or Early Termination
Description: as for outcome 7
Time Frame: Pre-dose on Day 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL
  IL-1alpha | 0.70 (0.68) | 0.66 (0.66)
  IL-1beta | 0.43 (0.43) | 0.38 (0.41)
  IL-4 | 0.29 (0.31) | 0.14 (0.13)
  IL-6 | 0.81 (0.46) | 0.66 (0.44)
  IL-7 | 0.85 (0.31) | 0.52 (0.35)
  IL-8 | 1.08 (0.26) | 1.04 (0.23)
  IL-10 | 0.22 (0.17) | 0.34 (0.37)
  IL-12p70 | 0.32 (0.26) | 0.33 (0.45)
  IL-17A | 0.43 (0.48) | 0.36 (0.35)
  IL-21 | 1.41 (1.04) | 1.58 (0.99)
  IP-10 | 2.20 (0.27) | 2.28 (0.38)
  TNFalpha | 0.46 (0.48) | 0.43 (0.51)
  IFNgamma | 0.17 (0.22) | 0.10 (0.00)
  G-CSF | 0.57 (0.55) | 0.58 (0.28)
  GM-CSF | 0.45 (0.46) | 0.35 (0.42)
  MCP1 | 2.17 (0.26) | 2.07 (0.35)
  MIP1a | 0.82 (0.50) | 0.85 (0.31)
  sVEGF | 1.92 (0.42) | 1.88 (0.29)
  sVCAM-1 | 4.97 (0.13) | 5.05 (0.16)
  sICAM-1 | 4.65 (0.12) | 4.76 (0.15)

16. Primary Outcome: Blood T, B and NK Lymphocyte Counts at Pre-dose on Day 1
Description: Blood samples were collected for fluorescence-activated cell sorting [FACS] analysis of lymphocyte subsets. Lymphocyte subset counts of T cells, Bone-marrow cells (B cells) and natural killer (NK) cells were analyzed using fluorescent-labeled antibodies against clusters of differentiation (CD) markers.
Time Frame: Pre-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells per microliter (cells/mcL)
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 11 | 12
cells per microliter (cells/mcL)
  B Cells (CD19) | 214.09 (134.72) | 389.17 (190.27)
  Total T Cells (CD3) | 1516.27 (567.38) | 1579.00 (628.89)
  CD8 T Cells (CD3 CD8) | 402.73 (205.74) | 376.67 (189.14)
  CD4 T Cells (CD3 CD4) | 1114.82 (415.59) | 1199.17 (496.66)
  NK Cells (CD16 CD56) | 276.45 (134.62) | 190.67 (121.20)
  Immature B Cells | 10.27 (11.23) | 8.83 (5.65)
  Naive Cells | 165.64 (113.99) | 273.67 (178.51)
  Marginal B Cells | 17.55 (7.62) | 81.50 (168.29)
  Memory B Cells | 20.45 (12.36) | 25.00 (14.83)
  Central Memory CD4 Cells | 627.45 (306.86) | 673.33 (291.75)
  Effector Memory CD4 Cells | 130.09 (138.98) | 93.92 (97.30)
  Naive CD4 Cells | 311.09 (245.67) | 420.92 (294.76)
  Terminally Differentiated(Diff) EffectorCD4 Cells | 45.82 (83.60) | 10.25 (15.15)
  Central Memory CD8 Cells | 117.73 (102.47) | 136.58 (77.79)
  Effector Memory CD8 Cells | 38.55 (29.88) | 68.25 (88.65)
  Naive CD8 Cells | 111.91 (81.86) | 113.08 (50.56)
  Terminally Diff Effector Memory CD8 Cells | 134.36 (140.97) | 58.83 (52.87)
  CD4 T-Cells | 81.91 (34.76) | 81.92 (42.95)
  CD56 Bright NK-Cells | 9.27 (3.85) | 7.00 (4.13)
  CD56 Dim NK-Cell | 209.09 (124.61) | 143.83 (103.97)
  CD56 Null NK-Cells | 57.82 (61.05) | 39.58 (27.28)
  CD56 Dim Null NK-Cells | 266.73 (132.17) | 183.42 (118.39)

17. Primary Outcome: Blood T, B and NK Lymphocyte Counts at 1 Hour Post-dose on Day 1
Description: Blood samples were collected for FACS analysis of lymphocyte subsets. Lymphocyte subset counts of T cells, B cells and NK cells were analyzed using fluorescent-labeled antibodies against CD markers.
Time Frame: 1 Hour Post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
cells/mcL
  B Cells (CD19) | 207.07 (128.57) | 312.69 (216.36)
  Total T Cells (CD3) | 1533.53 (631.42) | 1596.54 (754.87)
  CD8 T Cells (CD3 CD8) | 431.07 (229.21) | 372.38 (157.96)
  CD4 T Cells (CD3 CD4) | 1102.60 (450.53) | 1208.08 (651.25)
  NK Cells (CD16 CD56) | 422.87 (182.11) | 179.15 (107.03)
  Immature B Cells | 8.40 (9.63) | 8.92 (7.49)
  Naive Cells | 166.60 (111.95) | 222.75 (185.92)
  Marginal B Cells | 16.20 (6.65) | 78.17 (151.67)
  Memory B Cells | 16.07 (8.04) | 25.75 (17.78)
  Central Memory CD4 Cells | 640.07 (314.78) | 706.42 (360.34)
  Effector Memory CD4 Cells | 121.07 (127.98) | 61.83 (45.05)
  Naive CD4 Cells | 298.47 (197.32) | 459.75 (382.27)
  Terminally Diff Effector CD4 Cells | 42.93 (87.65) | 4.50 (6.78)
  Central Memory CD8 Cells | 134.40 (102.91) | 141.75 (87.65)
  Effector Memory CD8 Cells | 49.00 (37.44) | 46.58 (64.47)
  Naive CD8 Cells | 114.20 (50.74) | 137.33 (69.67)
  Terminally Diff Effector Memory CD8 Cells | 133.53 (168.92) | 39.58 (36.34)
  CD4 T-Cells | 76.13 (39.65) | 91.92 (55.68)
  CD56 Bright NK-Cells | 10.00 (4.75) | 7.23 (4.38)
  CD56 Dim NK-Cell | 358.33 (171.65) | 136.92 (97.23)
  CD56 Null NK-Cells | 54.40 (44.65) | 34.77 (23.81)
  CD56 Dim Null NK-Cells | 412.60 (180.18) | 171.62 (104.39)

18. Primary Outcome: Blood T, B and NK Lymphocyte Counts at 4 Hours Post-dose on Day 1
Description: as for outcome 17
Time Frame: 4 Hours Post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 12
cells/mcL
  B Cells (CD19) | 222.79 (154.52) | 380.33 (220.41)
  Total T Cells (CD3) | 1841.07 (880.14) | 1710.42 (959.80)
  CD8 T Cells (CD3 CD8) | 505.64 (298.97) | 393.00 (205.06)
  CD4 T Cells (CD3 CD4) | 1338.79 (633.15) | 1312.92 (834.04)
  NK Cells (CD16 CD56) | 428.50 (207.39) | 201.83 (192.98)
  Immature B Cells | 8.29 (10.41) | 10.92 (10.09)
  Naive Cells | 177.50 (129.90) | 265.00 (209.57)
  Marginal B Cells | 19.86 (12.60) | 74.83 (129.24)
  Memory B Cells | 17.07 (10.98) | 29.17 (23.94)
  Central Memory CD4 Cells | 785.43 (388.64) | 720.50 (383.62)
  Effector Memory CD4 Cells | 155.71 (165.49) | 93.42 (129.36)
  Naive CD4 Cells | 352.43 (307.49) | 488.75 (499.88)
  Terminally Diff Effector CD4 Cells | 45.57 (103.39) | 10.42 (18.37)
  Central Memory CD8 Cells | 159.21 (119.89) | 140.42 (90.69)
  Effector Memory CD8 Cells | 64.07 (52.87) | 61.33 (104.75)
  Naive CD8 Cells | 127.71 (54.79) | 142.42 (69.46)
  Terminally Diff Effector Memory CD8 Cells | 154.43 (201.13) | 48.67 (58.85)
  CD4 T-Cells | 86.36 (42.89) | 97.83 (78.84)
  CD56 Bright NK-Cells | 11.21 (6.05) | 7.17 (3.95)
  CD56 Dim NK-Cell | 364.57 (191.50) | 157.17 (158.85)
  CD56 Null NK-Cells | 52.57 (48.32) | 37.33 (37.57)
  CD56 Dim Null NK-Cells | 417.00 (204.21) | 194.50 (191.68)

19. Primary Outcome: Blood T, B and NK Lymphocyte Counts at Pre-dose on Day 10
Description: as for outcome 17
Time Frame: Pre-dose on Day 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 13
cells/mcL
  B Cells (CD19) | 290.50 (144.94) | 310.92 (154.13)
  Total T Cells (CD3) | 1732.29 (581.98) | 1477.08 (696.45)
  CD8 T Cells (CD3 CD8) | 413.64 (169.81) | 384.15 (216.57)
  CD4 T Cells (CD3 CD4) | 1314.64 (475.64) | 1084.62 (547.23)
  NK Cells (CD16 CD56) | 258.79 (177.98) | 205.38 (138.20)
  Immature B Cells | 11.21 (9.96) | 8.85 (7.99)
  Naive Cells | 218.57 (121.71) | 211.38 (133.45)
  Marginal B Cells | 32.29 (20.28) | 69.23 (135.70)
  Memory B Cells | 28.50 (14.53) | 21.31 (13.01)
  Central Memory CD4 Cells | 696.21 (294.16) | 603.54 (300.56)
  Effector Memory CD4 Cells | 130.86 (139.79) | 78.92 (102.26)
  Naive CD4 Cells | 453.86 (314.82) | 393.08 (296.88)
  Terminally Diff Effector CD4 Cells | 33.43 (52.47) | 9.31 (18.40)
  Central Memory CD8 Cells | 126.71 (95.74) | 132.46 (76.09)
  Effector Memory CD8 Cells | 37.57 (27.11) | 69.38 (104.84)
  Naive CD8 Cells | 136.93 (66.75) | 122.54 (91.92)
  Terminally Diff Effector Memory CD8 Cells | 112.50 (114.14) | 59.77 (70.15)
  CD4 T-Cells | 93.64 (57.44) | 79.69 (43.04)
  CD56 Bright NK-Cells | 5.07 (2.37) | 8.23 (4.80)
  CD56 Dim NK-Cell | 207.50 (162.82) | 149.54 (115.63)
  CD56 Null NK-Cells | 46.29 (52.45) | 47.46 (35.83)
  CD56 Dim Null NK-Cells | 253.64 (176.82) | 196.92 (136.36)

20. Primary Outcome: Blood T, B and NK Lymphocyte Counts at Pre-dose on Day 28
Description: as for outcome 17
Time Frame: Pre-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 12
cells/mcL
  B Cells (CD19) | 399.62 (208.61) | 392.25 (235.63)
  Total T Cells(CD3) | 1730.38 (730.18) | 1451.92 (622.86)
  CD8 T Cells (CD3 CD8) | 363.85 (143.45) | 346.58 (206.22)
  CD4 T Cells (CD3 CD4) | 1352.46 (618.78) | 1102.08 (454.72)
  NK Cells (CD16 CD56) | 184.92 (103.73) | 180.33 (123.31)
  Immature B Cells | 13.85 (8.99) | 11.25 (11.86)
  Naive Cells | 304.77 (177.06) | 280.50 (212.30)
  Marginal B Cells | 44.31 (36.38) | 73.75 (159.25)
  Memory B Cells | 36.69 (18.14) | 26.50 (19.50)
  Central Memory CD4 Cells | 736.00 (272.68) | 623.67 (259.72)
  Effector Memory CD4 Cells | 118.54 (91.20) | 90.00 (98.80)
  Naive CD4 Cells | 475.23 (421.51) | 378.50 (193.71)
  Terminally Diff Effector CD4 Cells | 22.69 (28.46) | 9.50 (14.13)
  Central Memory CD8 Cells | 120.69 (65.03) | 120.50 (68.09)
  Effector Memory CD8 Cells | 32.92 (25.69) | 55.50 (67.08)
  Naive CD8 Cells | 131.38 (85.53) | 121.75 (86.96)
  Terminally Diff Effector Memory CD8 Cells | 78.46 (81.53) | 49.00 (61.65)
  CD4 T-Cells | 84.38 (54.71) | 75.08 (43.97)
  CD56 Bright NK-Cells | 4.15 (2.03) | 7.17 (4.41)
  CD56 Dim NK-Cell | 127.15 (78.63) | 134.25 (103.99)
  CD56 Null NK-Cells | 53.77 (51.21) | 38.83 (35.54)
  CD56 Dim Null NK-Cells | 180.77 (103.02) | 173.17 (119.76)

21. Primary Outcome: Blood T, B and NK Lymphocyte Counts at 1 Hour Post-dose on Day 28
Description: as for outcome 17
Time Frame: 1 Hour Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
cells/mcL
  B Cells (CD19) | 343.21 (159.97) | 329.00 (202.97)
  Total T Cells(CD3) | 1705.57 (621.55) | 1630.64 (816.41)
  CD8 T Cells (CD3 CD8) | 409.71 (158.79) | 482.07 (388.11)
  CD4 T Cells (CD3 CD4) | 1281.00 (491.92) | 1145.50 (522.79)
  NK Cells (CD16 CD56) | 309.43 (112.95) | 339.50 (426.91)
  Immature B Cells | 12.43 (7.84) | 9.14 (9.04)
  Naive Cells | 261.57 (140.28) | 233.86 (171.68)
  Marginal B Cells | 36.43 (20.14) | 63.00 (141.24)
  Memory B Cells | 32.57 (15.27) | 23.07 (17.84)
  Central Memory CD4 Cells | 723.43 (253.15) | 614.50 (219.76)
  Effector Memory CD4 Cells | 117.21 (99.96) | 143.14 (237.16)
  Naive CD4 Cells | 418.93 (321.41) | 370.43 (199.66)
  Terminally Diff Effector CD4 Cells | 21.07 (31.32) | 17.43 (36.50)
  Central Memory CD8 Cells | 141.50 (82.12) | 128.14 (70.76)
  Effector Memory CD8 Cells | 36.07 (23.82) | 114.79 (187.14)
  Naive CD8 Cells | 135.29 (83.65) | 140.07 (101.82)
  Terminally Diff Effector Memory CD8 Cells | 97.21 (109.27) | 98.93 (154.16)
  CD4 T-Cells | 88.50 (51.93) | 78.64 (41.50)
  CD56 Bright NK-Cells | 4.71 (2.43) | 8.14 (5.53)
  CD56 Dim NK-Cell | 258.43 (111.98) | 284.14 (394.73)
  CD56 Null NK-Cells | 46.29 (25.38) | 46.93 (52.57)
  CD56 Dim Null NK-Cells | 304.64 (112.88) | 331.14 (422.93)

22. Primary Outcome: Blood T, B and NK Lymphocyte Counts at 4 Hours Post-dose on Day 28
Description: as for outcome 17
Time Frame: 4 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 11 | 12
cells/mcL
  B Cells (CD19) | 336.45 (194.70) | 347.67 (233.30)
  Total T Cells(CD3) | 1483.00 (495.98) | 1445.83 (712.35)
  CD8 T Cells (CD3 CD8) | 355.27 (111.71) | 346.00 (209.68)
  CD4 T Cells (CD3 CD4) | 1122.91 (419.02) | 1095.00 (565.70)
  NK Cells (CD16 CD56) | 188.36 (59.25) | 200.75 (191.26)
  Immature B Cells | 10.73 (8.33) | 10.33 (10.82)
  Naive Cells | 256.91 (156.81) | 247.17 (207.69)
  Marginal B Cells | 38.73 (38.69) | 67.17 (129.67)
  Memory B Cells | 29.91 (17.27) | 23.17 (19.64)
  Central Memory CD4 Cells | 675.55 (270.78) | 631.50 (260.76)
  Effector Memory CD4 Cells | 110.09 (69.34) | 85.92 (134.06)
  Naive CD4 Cells | 312.00 (237.45) | 369.50 (314.06)
  Terminally Diff Effector CD4 Cells | 24.91 (30.27) | 8.17 (20.56)
  Central Memory CD8 Cells | 118.09 (78.61) | 112.83 (60.76)
  Effector Memory CD8 Cells | 37.09 (27.50) | 60.17 (91.98)
  Naive CD8 Cells | 126.00 (90.18) | 133.17 (98.02)
  Terminally Diff Effector Memory CD8 Cells | 73.91 (58.79) | 40.00 (75.37)
  CD4 T-Cells | 64.09 (33.05) | 65.36 (36.70)
  CD56 Bright NK-Cells | 4.55 (2.42) | 6.83 (4.71)
  CD56 Dim NK-Cell | 143.55 (49.57) | 163.50 (158.10)
  CD56 Null NK-Cells | 40.36 (25.74) | 30.50 (35.48)
  CD56 Dim Null NK-Cells | 183.64 (58.53) | 193.92 (188.21)

23. Primary Outcome: Blood T, B and NK Lymphocyte Counts at 8 Hours Post-dose on Day 28
Description: as for outcome 17
Time Frame: 8 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 12 | 11
cells/mcL
  B Cells (CD19) | 382.33 (204.55) | 318.27 (253.87)
  Total T Cells(CD3) | 1557.58 (601.36) | 1616.00 (934.75)
  CD8 T Cells (CD3 CD8) | 348.33 (135.33) | 420.18 (226.60)
  CD4 T Cells (CD3 CD4) | 1203.67 (491.02) | 1186.73 (788.19)
  NK Cells (CD16 CD56) | 174.58 (82.07) | 217.91 (148.22)
  Immature B Cells | 11.25 (7.10) | 7.30 (8.08)
  Naive Cells | 291.33 (165.84) | 243.10 (220.30)
  Marginal B Cells | 46.50 (38.57) | 76.60 (142.34)
  Memory B Cells | 33.00 (20.82) | 22.70 (19.96)
  Central Memory CD4 Cells | 726.75 (293.12) | 725.00 (424.16)
  Effector Memory CD4 Cells | 119.17 (87.92) | 85.64 (127.90)
  Naive CD4 Cells | 338.17 (270.26) | 367.73 (378.39)
  Terminally Diff Effector CD4 Cells | 19.83 (21.41) | 8.27 (18.79)
  Central Memory CD8 Cells | 115.92 (51.47) | 149.27 (86.30)
  Effector Memory CD8 Cells | 35.33 (25.27) | 85.09 (110.75)
  Naive CD8 Cells | 133.25 (95.54) | 133.64 (111.11)
  Terminally Diff Effector Memory CD8 Cells | 64.08 (56.47) | 52.27 (72.48)
  CD4 T-Cells | 79.00 (53.92) | 89.50 (72.98)
  CD56 Bright NK-Cells | 3.36 (1.80) | 7.27 (4.29)
  CD56 Dim NK-Cell | 117.18 (59.33) | 164.36 (125.72)
  CD56 Null NK-Cells | 41.91 (29.36) | 46.27 (38.40)
  CD56 Dim Null NK-Cells | 158.91 (74.78) | 210.64 (145.85)

24. Primary Outcome: Blood T, B and NK Lymphocyte Counts at 24 Hours Post-dose on Day 28
Description: as for outcome 17
Time Frame: 24 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 12 | 12
cells/mcL
  B Cells (CD19) | 276.00 (167.25) | 300.92 (191.57)
  Total T Cells(CD3) | 1044.08 (505.60) | 1619.33 (913.77)
  CD8 T Cells (CD3 CD8) | 239.92 (113.32) | 382.75 (200.38)
  CD4 T Cells (CD3 CD4) | 799.50 (408.07) | 1223.17 (779.67)
  NK Cells (CD16 CD56) | 92.92 (52.30) | 196.67 (152.83)
  Immature B Cells | 10.00 (4.20) | 9.75 (9.52)
  Naive Cells | 215.83 (146.07) | 245.33 (173.16)
  Marginal B Cells | 25.58 (18.78) | 24.08 (27.05)
  Memory B Cells | 24.83 (11.10) | 21.75 (16.10)
  Central Memory CD4 Cells | 431.92 (186.89) | 626.00 (339.12)
  Effector Memory CD4 Cells | 59.58 (41.84) | 79.50 (119.68)
  Naive CD4 Cells | 297.17 (287.44) | 508.83 (483.29)
  Terminally Diff Effector CD4 Cells | 11.00 (18.39) | 9.00 (18.01)
  Central Memory CD8 Cells | 85.50 (72.10) | 133.33 (83.39)
  Effector Memory CD8 Cells | 16.75 (8.58) | 59.17 (93.93)
  Naive CD8 Cells | 89.25 (62.57) | 142.08 (131.13)
  Terminally Diff Effector Memory CD8 Cells | 48.42 (55.68) | 48.17 (60.46)
  CD4 T Cells | 61.67 (41.32) | 92.58 (59.44)
  CD56 Bright NK-Cells | 1.83 (1.11) | 8.50 (4.76)
  CD56 Dim NK-Cell | 65.42 (47.76) | 158.17 (137.82)
  CD56 Null NK-Cells | 25.50 (12.72) | 30.08 (26.57)
  CD56 Dim Null NK-Cells | 91.08 (51.61) | 187.92 (149.63)

25. Primary Outcome: Blood T, B and NK Lymphocyte Counts and Possible Subsets at Pre-dose on Day 35 or Early Termination
Description: as for outcome 17
Time Frame: Pre-dose on Day 35 or Early Termination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 12
cells/mcL
  B Cells (CD19) | 173.86 (95.29) | 344.17 (211.00)
  Total T Cells (CD3) | 1044.07 (529.37) | 1411.75 (474.97)
  CD8 T Cells (CD3+CD8) | 253.64 (190.57) | 364.92 (202.70)
  CD4 T Cells (CD3 CD4) | 781.57 (350.40) | 1046.00 (328.08)
  NK Cells (CD16 CD56) | 162.21 (116.20) | 179.67 (142.64)
  Immature B Cells | 5.57 (3.59) | 11.17 (9.99)
  Naive Cells | 136.43 (80.37) | 252.92 (206.67)
  Marginal B Cells | 15.50 (8.72) | 57.58 (102.20)
  Memory B Cells | 16.36 (12.73) | 22.50 (13.93)
  Central Memory CD4 Cells | 416.93 (167.72) | 605.00 (222.14)
  Effector Memory CD4 Cells | 56.29 (51.24) | 97.25 (103.24)
  Naive CD4 Cells | 290.36 (244.79) | 333.83 (132.59)
  Terminally Diff Effector CD4 Cells | 18.00 (24.88) | 9.75 (16.44)
  Central Memory CD8 Cells | 73.71 (58.46) | 109.42 (49.90)
  Effector Memory CD8 Cells | 17.93 (13.74) | 70.58 (99.36)
  Naive CD8 Cells | 101.79 (126.51) | 133.75 (97.93)
  Terminally Diff Effector Memory CD8 Cells | 60.07 (67.10) | 51.08 (61.27)
  CD4 T Cells | 66.64 (40.58) | 73.50 (39.02)
  CD56 Bright NK-Cells | 3.62 (2.60) | 6.33 (3.52)
  CD56 Dim NK-Cell | 99.00 (89.92) | 141.17 (130.25)
  CD56 Null NK-Cells | 66.23 (72.59) | 32.25 (19.30)
  CD56 Dim Null NK-Cells | 165.15 (115.88) | 173.25 (141.06)

26. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at Pre-dose on Day 1
Description: Blood/serum samples were analyzed for MMP3, osteocalcin and osteopontin concentrations using a validated analytical assay sensitive and specific Enzyme-Linked Immunosorbent Assay [ELISA] method for MMP3 and osteopontin in serum samples; specific electrochemiluminescence method for osteocalcin in blood samples).
Time Frame: Pre-dose on Day 1
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
nanogram per milliliter (ng/mL)
  MMP3 | 38.31 (32.24) | 24.52 (12.65)
  Osteocalcin | 19.54 (8.23) | 18.54 (12.31)
  Osteopontin | 108.40 (42.59) | 98.11 (37.04)

27. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at 1 Hour Post-dose on Day 1
Description: Blood/serum samples were analyzed for MMP3, osteocalcin and osteopontin concentrations using a validated analytical assay sensitive and specific ELISA method for MMP3 and osteopontin in serum samples; specific electrochemiluminescence method for osteocalcin in blood samples.
Time Frame: 1 Hour Post-dose on Day 1
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
ng/mL
  MMP3 | 37.30 (32.40) | 22.42 (12.06)
  Osteocalcin | 18.90 (8.12) | 18.01 (11.38)
  Osteopontin | 101.10 (40.23) | 94.37 (39.02)

28. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at 4 Hours Post-dose on Day 1
Description: as for outcome 27
Time Frame: 4 Hours Post-dose on Day 1
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
ng/mL
  MMP3 | 36.98 (30.72) | 22.09 (12.08)
  Osteocalcin | 18.17 (7.30) | 19.01 (13.17)
  Osteopontin | 99.82 (36.77) | 95.23 (38.37)

29. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at Pre-dose on Day 10
Description: as for outcome 27
Time Frame: Pre-dose on Day 10
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
ng/mL
  MMP3 | 32.10 (26.89) | 21.05 (12.28)
  Osteocalcin | 21.35 (8.87) | 18.60 (11.28)
  Osteopontin | 91.13 (29.16) | 91.12 (34.13)

30. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at Pre-dose on Day 28
Description: as for outcome 27
Time Frame: Pre-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
ng/mL
  MMP3 | 25.18 (22.33) | 19.26 (11.64)
  Osteocalcin | 22.05 (9.28) | 16.51 (9.06)
  Osteopontin | 78.23 (17.23) | 79.93 (18.63)

31. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at 1 Hour Post-dose on Day 28
Description: as for outcome 27
Time Frame: 1 Hour Post-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
ng/mL
  MMP3 | 21.59 (19.30) | 18.86 (11.73)
  Osteocalcin | 21.45 (9.65) | 17.37 (8.85)
  Osteopontin | 78.60 (19.24) | 86.66 (29.65)

32. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at 4 Hours Post-dose on Day 28
Description: as for outcome 27
Time Frame: 4 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 13
ng/mL
  MMP3 | 19.71 (17.65) | 16.67 (10.70)
  Osteocalcin | 21.09 (8.26) | 15.45 (7.22)
  Osteopontin | 71.52 (24.92) | 86.56 (33.00)

33. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at 8 Hours Post-dose on Day 28
Description: as for outcome 27
Time Frame: 8 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 12
ng/mL
  MMP3 | 17.94 (14.38) | 16.68 (11.75)
  Osteocalcin | 20.93 (6.37) | 16.67 (8.63)
  Osteopontin | 75.32 (21.32) | 89.84 (33.02)

34. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at 24 Hours Post-dose on Day 28
Description: as for outcome 27
Time Frame: 24 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
ng/mL
  MMP3 | 24.48 (20.82) | 26.20 (15.56)
  Osteocalcin | 20.96 (9.45) | 17.49 (9.57)
  Osteopontin | 82.60 (22.28) | 95.51 (28.50)

35. Primary Outcome: Matrix Metallopeptidase 3 (MMP3), Osteocalcin and Osteopontin Levels at Pre-dose on Day 35 or Early Termination
Description: as for outcome 27
Time Frame: Pre-dose on Day 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
ng/mL
  MMP3 | 28.98 (21.36) | 28.72 (24.48)
  Osteocalcin | 21.79 (9.38) | 16.60 (10.48)
  Osteopontin | 95.93 (29.73) | 86.48 (29.69)

36. Primary Outcome: Parathyroid Hormone (PTH) Level at Pre-dose on Day 1
Description: Plasma samples were analyzed for PTH concentrations using a validated, sensitive and specific electrochemiluminescence method.
Time Frame: Pre-dose on Day 1
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL | 38.40 (17.44) | 33.32 (5.80)

37. Primary Outcome: Parathyroid Hormone (PTH) Level at 1 Hour Post-dose on Day 1
Description: as for outcome 36
Time Frame: 1 Hour Post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
pg/mL | 33.89 (13.44) | 31.48 (8.77)

38. Primary Outcome: Parathyroid Hormone (PTH) Level at 4 Hours Post-dose on Day 1
Description: as for outcome 36
Time Frame: 4 Hours Post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 13
pg/mL | 32.97 (13.31) | 33.35 (7.12)

39. Primary Outcome: Parathyroid Hormone (PTH) Level at Pre-dose on Day 10
Description: as for outcome 36
Time Frame: Pre-dose on Day 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
pg/mL | 34.93 (11.76) | 31.48 (8.37)

40. Primary Outcome: Parathyroid Hormone (PTH) Level at Pre-dose on Day 28
Description: as for outcome 36
Time Frame: Pre-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
pg/mL | 38.46 (12.64) | 33.39 (8.94)

41. Primary Outcome: Parathyroid Hormone (PTH) Level at 1 Hour Post-dose on Day 28
Description: as for outcome 36
Time Frame: 1 Hour Post-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL | 37.97 (14.05) | 33.93 (7.51)

42. Primary Outcome: Parathyroid Hormone (PTH) Level at 4 Hours Post-dose on Day 28
Description: as for outcome 36
Time Frame: 4 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 13
pg/mL | 38.70 (13.25) | 36.65 (12.54)

43. Primary Outcome: Parathyroid Hormone (PTH) Level at 8 Hours Post-dose on Day 28
Description: as for outcome 36
Time Frame: 8 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 11
pg/mL | 37.76 (15.90) | 37.82 (18.84)

44. Primary Outcome: Parathyroid Hormone (PTH) Level at 24 Hours Post-dose on Day 28
Description: as for outcome 36
Time Frame: 24 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 12
pg/mL | 35.91 (19.94) | 36.08 (10.17)

45. Primary Outcome: Parathyroid Hormone (PTH) Level at Pre-dose on Day 35 or Early Termination
Description: as for outcome 36
Time Frame: Pre-dose on Day 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL | 37.30 (14.86) | 34.59 (10.40)

46. Primary Outcome: Osteoprotegerin (OPG) Level at Pre-dose on Day 1
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: Pre-dose on Day 1
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
picomole per liter (pmol/L) | 5.99 (2.04) | 6.21 (1.91)

47. Primary Outcome: Osteoprotegerin (OPG) Level at 1 Hour Post-dose on Day 1
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 1 Hour Post-dose on Day 1
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pmol/L | 6.13 (1.99) | 5.72 (2.16)

48. Primary Outcome: Osteoprotegerin (OPG) Level at 4 Hours Post-dose on Day 1
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 4 Hours Post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
picomole per liter (pmol/L) | 5.50 (1.53) | 5.35 (1.86)

49. Primary Outcome: Osteoprotegerin (OPG) Level at Pre-dose on Day 10
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: Pre-dose on Day 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
pmol/L | 6.02 (1.88) | 5.82 (2.22)

50. Primary Outcome: Osteoprotegerin (OPG) Level at Pre-dose on Day 28
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: Pre-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pmol/L | 5.53 (1.79) | 5.64 (2.48)

51. Primary Outcome: Osteoprotegerin (OPG) Level at 1 Hour Post-dose on Day 28
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 1 Hour Post-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pmol/L | 5.72 (1.86) | 5.56 (2.14)

52. Primary Outcome: Osteoprotegerin (OPG) Level at 4 Hours Post-dose on Day 28
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 4 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 13
pmol/L | 5.18 (1.55) | 5.69 (2.13)

53. Primary Outcome: Osteoprotegerin (OPG) Level at 8 Hours Post-dose on Day 28
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 8 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 12
pmol/L | 4.64 (1.28) | 5.64 (2.39)

54. Primary Outcome: Osteoprotegerin (OPG) Level at 24 Hours Post-dose on Day 28
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 24 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
pmol/L | 7.22 (2.74) | 6.20 (2.07)

55. Primary Outcome: Osteoprotegerin(OPG) Level at Pre-dose on Day 35 or Early Termination
Description: Blood samples were analyzed for OPG concentrations using a validated, sensitive and specific ELISA method.
Time Frame: Pre-dose on Day 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pmol/L | 6.31 (1.70) | 5.65 (2.01)

56. Primary Outcome: Plasma Level of Matrix Metallopeptidase (MMP13)
Time Frame: Pre-dose on Day 1, 10, 28 and 35 or Early Termination; 1, 4 hours Post-dose on Day 1, 28; 8, 24 hours Post-dose on Day 28
Population: Analyses of MMP13 was not performed as valid assay for MMP13 was not available.
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 0 | 0

57. Primary Outcome: Plasma Level of Interleukin-34 (IL-34) and Interleukin-18 (IL-18)
Time Frame: as for outcome 56
Population: Analyses of IL-34 and IL-18 were not performed as a valid assay was not available.
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 0 | 0

58. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at Pre-dose on Day 1
Description: Serum samples were analyzed for SAA concentrations using meso scale discovery (MSD) single ELISA electrochemiluminescence method and for CTX-1 concentrations using a validated, sensitive and specific Electro ChemiLuminescent ImmunoAssay (ECLIA).
Time Frame: Pre-dose on Day 1
Population: FAS included all randomized participants who received at least 1 dose of the study medication. Here, 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure. n=participants evaluable for this measure at specified time points for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
ng/mL
  SAA (n=14, 14) | 26383.03 (43196.37) | 23427.00 (43431.26)
  CTX-1 (n=14, 12) | 0.43 (0.26) | 0.37 (0.27)

59. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at 1 Hour Post-dose on Day 1
Description: Serum samples were analyzed for SAA concentrations using MSD single ELISA electrochemiluminescence method and for CTX-1 concentrations using a validated, sensitive and specific ECLIA.
Time Frame: 1 Hour Post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
ng/mL
  SAA | 25716.93 (42986.70) | 23308.57 (41911.51)
  CTX-1 | 0.36 (0.25) | 0.32 (0.22)

60. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at 4 Hours Post-dose on Day 1
Description: as for outcome 59
Time Frame: 4 Hours Post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 13
ng/mL
  SAA | 26460.26 (46059.64) | 27297.36 (52346.36)
  CTX-1 | 0.25 (0.12) | 0.25 (0.19)

61. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at Pre-dose on Day 10
Description: as for outcome 59
Time Frame: Pre-dose on Day 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
ng/mL
  SAA | 5968.89 (5509.18) | 31666.50 (92833.52)
  CTX-1 | 0.34 (0.16) | 0.35 (0.22)

62. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at Pre-dose on Day 28
Description: as for outcome 59
Time Frame: Pre-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
ng/mL
  SAA | 4094.94 (2527.72) | 14818.88 (18346.19)
  CTX-1 | 0.36 (0.19) | 0.35 (0.19)

63. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at 1 Hour Post-dose on Day 28
Description: as for outcome 59
Time Frame: 1 Hour Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
ng/mL
  SAA | 3921.49 (2291.33) | 18976.74 (29228.65)
  CTX-1 | 0.32 (0.16) | 0.35 (0.25)

64. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at 4 Hours Post-dose on Day 28
Description: as for outcome 59
Time Frame: 4 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 13
ng/mL
  SAA | 4042.21 (2974.03) | 20123.97 (31463.56)
  CTX-1 | 0.29 (0.17) | 0.20 (0.12)

65. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at 8 Hours Post-dose on Day 28
Description: as for outcome 59
Time Frame: 8 Hours Post-dose on Day 28
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 12
ng/mL
  SAA (n=14, 12) | 4113.05 (2939.86) | 15403.08 (24616.14)
  CTX-1 (n=12, 12) | 0.28 (0.17) | 0.31 (0.21)

66. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at 24 Hours Post-dose on Day 28
Description: as for outcome 59
Time Frame: 24 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 14
ng/mL
  SAA | 6643.14 (6504.55) | 14627.28 (16685.62)
  CTX-1 | 0.28 (0.16) | 0.28 (0.13)

67. Primary Outcome: Serum Amyloid A (SAA) and Carboxy-Terminal Collagen Crosslinks-1 (CTX-1) Levels at Pre-dose on Day 35 or Early Termination
Description: as for outcome 59
Time Frame: Pre-dose on Day 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
ng/mL
  SAA | 22174.19 (25387.79) | 33853.61 (88542.43)
  CTX-1 | 0.27 (0.15) | 0.34 (0.16)

68. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at Pre-dose on Day 1
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: Pre-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 13
pg/mL
  IL-1ra | 545.71 (279.48) | 449.38 (163.85)
  IL-15 | 8.00 (0.00) | 8.00 (0.00)

69. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at 1 Hour Post-dose on Day 1
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 1 Hour Post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
pg/mL
  IL-1ra | 565.43 (262.73) | 479.93 (167.61)
  IL-15 | 8.00 (0.00) | 8.00 (0.00)

70. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at 4 Hours Post-dose on Day 1
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 4 Hours Post-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 13
pg/mL
  IL-1ra | 518.29 (297.33) | 477.25 (142.17)
  IL-15 | 8.00 (0.00) | 8.00 (0.00)

71. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at Pre-dose on Day 10
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: Pre-dose on Day 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
pg/mL
  IL-1ra | 487.00 (265.16) | 465.00 (176.17)
  IL-15 | 8.00 (0.00) | 8.00 (0.00)

72. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at Pre-dose on Day 28
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: Pre-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
pg/mL
  IL-1ra | 437.73 (171.93) | 617.38 (624.81)
  IL-15 | 8.00 (0.00) | 8.00 (0.00)

73. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at 1 Hour Post-dose on Day 28
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 1 Hour Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 13
pg/mL
  IL-1ra | 421.00 (196.57) | 501.31 (337.85)
  IL-15 | 8.00 (0.00) | 8.00 (0.00)

74. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at 4 Hours Post-dose on Day 28
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 4 Hours Post-dose on Day 28
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 13
pg/mL
  IL-1ra (n= 13, 13) | 388.15 (147.27) | 552.85 (415.32)
  IL-15 (n=11, 12) | 8.00 (0.00) | 8.00 (0.00)

75. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at 8 Hours Post-dose on Day 28
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 8 Hours Post-dose on Day 28
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 12 | 12
pg/mL
  IL-1ra (n=12, 12) | 399.08 (157.84) | 414.67 (152.99)
  IL-15 (n=12, 10) | 8.00 (0.00) | 8.00 (0.00)

76. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at 24 Hours Post-dose on Day 28
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: 24 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 14
pg/mL
  IL-1ra | 500.38 (187.55) | 462.57 (175.80)
  IL-15 | 8.26 (0.94) | 8.00 (0.00)

77. Primary Outcome: Interleukin-1 Receptor Antagonist (IL-1ra) and Interleukin-15 (IL-15) Levels at Pre-dose on Day 35 or Early Termination
Description: Serum samples were analyzed for IL-1ra and IL-15 concentrations using a validated, sensitive and specific ELISA method.
Time Frame: Pre-dose on Day 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
pg/mL
  IL-1ra | 520.87 (282.88) | 486.57 (317.27)
  IL-15 | 8.00 (0.00) | 8.00 (0.00)

78. Primary Outcome: Urine Collagen Type II C-telopeptide Fragments (uCTX-II) at Pre-dose on Day 1
Description: Urinary concentration of collagen type II C-telopeptide fragments was measured by competitive ELISA. uCTX-II was measured as nanogram per millimoles of creatinine (ng/mmol Cr).
Time Frame: Pre-dose on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mmol Cr
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 13 | 13
ng/mmol Cr | 454.74 (216.74) | 345.87 (259.83)

79. Primary Outcome: Urine Collagen Type II C-telopeptide Fragments (uCTX-II) at Pre-dose on Day 10
Description: Urinary concentration of collagen type II C-telopeptide fragments was measured by competitive ELISA. uCTX-II was measured as ng/mmol Cr.
Time Frame: Pre-dose on Day 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mmol Cr
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
ng/mmol Cr | 318.10 (208.07) | 423.76 (389.15)

80. Primary Outcome: Urine Collagen Type II C-telopeptide Fragments (uCTX-II) at Pre-dose on Day 28
Description: as for outcome 79
Time Frame: Pre-dose on Day 28
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: ng/mmol Cr
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
ng/mmol Cr | 320.42 (192.31) | 409.89 (338.67)

81. Primary Outcome: Urine Collagen Type II C-telopeptide Fragments (uCTX-II) at 24 Hours Post-dose on Day 28
Description: as for outcome 79
Time Frame: 24 Hours Post-dose on Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mmol Cr
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 13
ng/mmol Cr | 267.86 (159.63) | 284.87 (202.92)

82. Primary Outcome: Urine Collagen Type II C-telopeptide Fragments (uCTX-II) at Pre-dose on Day 35 or Early Termination
Description: as for outcome 79
Time Frame: Pre-dose on Day 35 or Early Termination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mmol Cr
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 14 | 14
ng/mmol Cr | 278.55 (198.90) | 340.83 (379.42)

83. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% Response
Description: ACR20 response: greater than or equal to (>=) 20 percent (%) improvement in tender joint count (TJC); >= 20% improvement in swollen joint count (SJC); and >= 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Day 28, 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
percentage of participants
  Day 28 | 60.0 | 0.0
  Day 35 or Early Termination | 33.3 | 0.0

84. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: >=50% improvement in TJC; >= 50% improvement in SJC; and 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Day 28, 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
percentage of participants
  Day 28 | 40.0 | 0.0
  Day 35 or Early Termination | 13.3 | 0.0

85. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: >=70% improvement in TJC; >= 70% improvement in SJC; and 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Day 28, 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
percentage of participants
  Day 28 | 6.7 | 0.0
  Day 35 or Early Termination | 6.7 | 0.0

86. Secondary Outcome: Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP])
Description: DAS28-3 (CRP) was calculated from the SJC, TJC using the 28 joints count and the CRP) (milligram per liter [mg/L]). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) less than or equal to (<=) 3.2 implied low disease activity, greater than (>) 3.2 to 5.1 implied moderate to high disease activity and less than (<) 2.6 implied remission.
Time Frame: Day -7, 1 (Baseline), 28, 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
units on a scale
  Day -7 | 5.58 (0.87) | 5.06 (1.16)
  Day 1 (Baseline) | 5.57 (0.78) | 5.22 (0.96)
  Day 28 | 4.06 (0.97) | 4.91 (0.92)
  Day 35 or Early Termination | 4.91 (1.10) | 4.79 (1.10)

87. Secondary Outcome: Change From Baseline in Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Day 28 and 35
Description: DAS28-3 (CRP) was calculated from the SJC, TJC using the 28 joints count and the CRP (mg/mL). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-3 (CRP) <= 3.2 implied low disease activity, >3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Day 1 (Baseline), 28, 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
units on a scale
  Day 28 | -1.51 (0.97) | -0.31 (0.49)
  Day 35 or Early Termination | -0.66 (0.96) | -0.43 (0.40)

88. Secondary Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) <=3.2 and <2.6
Description: as for outcome 87
Time Frame: Day -7, 1 (Baseline), 28, 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
percentage of participants
  Day -7: DAS28-3 (CRP) <=3.2 | 0.0 | 7.1
  Day -7: DAS28-3 (CRP) <2.6 | 0.0 | 0.0
  Day 1 (Baseline): DAS28-3 (CRP) <=3.2 | 0.0 | 0.0
  Day 1 (Baseline): DAS28-3 (CRP) <2.6 | 0.0 | 0.0
  Day 28: DAS28-3 (CRP) <=3.2 | 20.0 | 14.3
  Day 28: DAS28-3 (CRP) <2.6 | 0.0 | 0.0
  Day 35 or Early Termination: DAS28-3 (CRP) <=3.2 | 6.7 | 7.1
  Day 35 or Early Termination: DAS28-3 (CRP) <2.6 | 0.0 | 0.0

89. Secondary Outcome: Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])
Description: DAS28-4 (ESR) was calculated from the number of SJC, TJC using the 28 joints count, ESR (millimeters per hour [mm/hour]) and patient's global assessment (PtGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity, > 3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Day -7, 1 (Baseline), 28, 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
units on a scale
  Day -7 | 6.60 (0.98) | 6.17 (1.12)
  Day 1 (Baseline) | 6.55 (0.98) | 6.32 (1.01)
  Day 28 | 4.90 (1.11) | 6.03 (0.98)
  Day 35 or Early Termination | 5.83 (1.23) | 6.00 (1.01)

90. Secondary Outcome: Change From Baseline in Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) at Day 28 and 35
Description: DAS28-4 (ESR) was calculated from the number of SJC, TJC using the 28 joints count, ESR [mm/hour] and patient's global assessment (PtGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). Total score range: 0 to 9.4, higher score indicated more disease activity. DAS28-4 (ESR) <= 3.2 implied low disease activity, > 3.2 to 5.1 implied moderate to high disease activity and <2.6 implied remission.
Time Frame: Day 1 (Baseline), 28, 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
units on a scale
  Day 28 | -1.58 (1.02) | -0.30 (0.60)
  Day 35 or Early Termination | -0.73 (0.91) | -0.32 (0.50)

91. Secondary Outcome: Percentage of Participants With Disease Activity Score Using 28-Joint Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR]) <=3.2 and <2.6
Description: as for outcome 90
Time Frame: Day -7, 1 (Baseline), 28, 35 or Early Termination
Population: FAS included all randomized participants who received at least 1 dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 | Placebo
Number analyzed (Participants) | 15 | 14
percentage of participants
  Day -7: DAS28-4 (ESR) =<3.2 | 0.0 | 0.0
  Day -7: DAS28-4 (ESR) <2.6 | 0.0 | 0.0
  Day 1 (Baseline): DAS28-4 (ESR) =<3.2 | 0.0 | 0.0
  Day 1 (Baseline): DAS28-4 (ESR) <2.6 | 0.0 | 0.0
  Day 28: DAS28-4 (ESR) =<3.2 | 7.1 | 0.0
  Day 28: DAS28-4 (ESR) <2.6 | 0.0 | 0.0
  Day 35 or Early Termination: DAS28-4 (ESR) =<3.2 | 0.0 | 0.0
  Day 35 or Early Termination: DAS28-4 (ESR) <2.6 | 0.0 | 0.0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | CP-690,550 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 7/15 | 10/14
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 (N=15) | Placebo (N=14)
Constipation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.